CLINICAL TRIAL: NCT05690412
Title: Efficacy and Safety of Endoscopic Papillectomy in the Treatment of Ampullary Neoplasms: a Multicenter, Retrospective, Nationwide Study.
Brief Title: Efficacy and Safety of Endoscopic Papillectomy in the Treatment of Ampullary Neoplasms.
Acronym: PaNETh
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Principal Investigator, Carlo Fabbri, Chief of Gastroenterology and Digestive Endoscopy Unit, Forlì-Cesena Hospitals, Azienda Unità Sanitaria Locale della Romagna
Other Study IDs: 2828
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Ampullary Adenoma; Ampulla of Vater Adenoma; Ampullary Cancer; Ampulla of Vater Cancer
Keywords: Endoscopic Papillectomy; Ampullary Adenoma; Ampullary Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Papillectomy — Endoscopic resection of ampullary neoplasm

SUMMARY:
The aim of our study is to provide data on the efficacy and safety of endoscopic papillectomy, by including consecutive patients treated after 2015, when first guidelines on endoscopic management of ampullary neoplasms were available.

DETAILED DESCRIPTION:
Ampullary neoplasm (AN) is a rare disease, but its incidence is increasing. In the last 20 years, endoscopic papillectomy (EP) has become the gold standard treatment for ampullary adenomas and early stage adenocarcinomas, thereby replacing surgical resection, which is burdened by higher rates of morbidity and mortality. However, the data supporting safety and efficacy of EP derive from multiple retrospective studies, that included procedures mostly performed before 2015, when first guidelines on endoscopic management of AN were available. This had an impact on large variability in patient selection criteria and endoscopic techniques, resulting in heterogenous outcomes. Therefore, the aim of our study is to provide data on the efficacy and safety of this technique, by including consecutive patients treated after the standardization of this technique.

All patients who underwent EP at 19 Italian centers between January 2016 and December 2021 were included. Clinical success was defined by the complete endoscopic management of the neoplasm and any eventual recurrence found in the follow-up period. EP-related adverse events and recurrences were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ampullary neoplasm, confirmed by histological examination of the endoscopically resected specimen

Exclusion Criteria:

* Absence of dysplasia on the resected specimen;
* Locally advanced or metastatic disease (Clinical TNM stage >T1 or N+ or M+);
* Neoplasm Intra-Ductal Extension (IDE) > 20 mm;
* Previously treated ampullary neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent Endoscopic Papillectomy for Ampullary Neoplasm at 19 Italian centers, between January 2016 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 2016-2021
  Complete endoscopic management of the neoplasm and any eventual recurrence found in the follow-up period.

SECONDARY OUTCOMES:
Adverse Events | 2016-2021
  Incidence of Endoscopic Papillectomy-related adverse events.
Recurrences | 2016-2021
  Incidence of neoplastic recurrences in the follow-up period, after Endoscopic Papillectomy.
Concordance between pre- and post-Endoscopic Papillectomy pathologic findings | 2016-2021
  Concordance between pre- and post-Endoscopic Papillectomy pathologic findings

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Morgagni-Pierantoni, Forlì, Forlì-Cesena, Italy

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Chathadi KV, Khashab MA, Acosta RD, Chandrasekhara V, Eloubeidi MA, Faulx AL, Fonkalsrud L, Lightdale JR, Salztman JR, Shaukat A, Wang A, Cash BD, DeWitt JM. The role of endoscopy in ampullary and duodenal adenomas. Gastrointest Endosc. 2015 Nov;82(5):773-81. doi: 10.1016/j.gie.2015.06.027. Epub 2015 Aug 7. No abstract available. PMID 26260385
- [Background] Vanbiervliet G, Strijker M, Arvanitakis M, Aelvoet A, Arnelo U, Beyna T, Busch O, Deprez PH, Kunovsky L, Larghi A, Manes G, Moss A, Napoleon B, Nayar M, Perez-Cuadrado-Robles E, Seewald S, Barthet M, van Hooft JE. Endoscopic management of ampullary tumors: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Apr;53(4):429-448. doi: 10.1055/a-1397-3198. Epub 2021 Mar 16. PMID 33728632
- [Background] Spadaccini M, Fugazza A, Frazzoni L, Leo MD, Auriemma F, Carrara S, Maselli R, Galtieri PA, Chandrasekar VT, Fuccio L, Aljahdli E, Hassan C, Sharma P, Anderloni A, Repici A. Endoscopic papillectomy for neoplastic ampullary lesions: A systematic review with pooled analysis. United European Gastroenterol J. 2020 Feb;8(1):44-51. doi: 10.1177/2050640619868367. Epub 2019 Jul 30. PMID 32213054
- [Background] Napoleon B, Gincul R, Ponchon T, Berthiller J, Escourrou J, Canard JM, Boyer J, Barthet M, Ponsot P, Laugier R, Helbert T, Coumaros D, Scoazec JY, Mion F, Saurin JC; Societe Francaise d'Endoscopie Digestive (SFED, French Society of Digestive Endoscopy). Endoscopic papillectomy for early ampullary tumors: long-term results from a large multicenter prospective study. Endoscopy. 2014 Feb;46(2):127-34. doi: 10.1055/s-0034-1364875. Epub 2014 Jan 29. PMID 24477368
- [Background] Tringali A, Valerii G, Boskoski I, Familiari P, Landi R, Perri V, Costamagna G. Endoscopic snare papillectomy for adenoma of the ampulla of vater: Long-term results in 135 consecutive patients. Dig Liver Dis. 2020 Sep;52(9):1033-1038. doi: 10.1016/j.dld.2020.05.029. Epub 2020 Jun 10. PMID 32532606
- [Background] Cecinato P, Parmeggiani F, Braglia L, Carlinfante G, Zecchini R, Decembrino F, Iori V, Sereni G, Tioli C, Cavina M, Camellini L, Azzolini F, Ponz de Leon M, Sassatelli R. Endoscopic Papillectomy for Ampullary Adenomas: Different Outcomes in Sporadic Tumors and Those Associated with Familial Adenomatous Polyposis. J Gastrointest Surg. 2021 Feb;25(2):457-466. doi: 10.1007/s11605-019-04500-w. Epub 2020 Jan 2. PMID 31898110
- [Background] Fritzsche JA, Klein A, Beekman MJ, van Hooft JE, Sidhu M, Schoeman S, Fockens P, Bourke MJ, Voermans RP. Endoscopic papillectomy; a retrospective international multicenter cohort study with long-term follow-up. Surg Endosc. 2021 Nov;35(11):6259-6267. doi: 10.1007/s00464-020-08126-x. Epub 2020 Nov 6. PMID 33159297
- [Background] Gondran H, Musquer N, Perez-Cuadrado-Robles E, Deprez PH, Buisson F, Berger A, Cesbron-Metivier E, Wallenhorst T, David N, Cholet F, Perrot B, Queneherve L, Coron E. Efficacy and safety of endoscopic papillectomy: a multicenter, retrospective, cohort study on 227 patients. Therap Adv Gastroenterol. 2022 Apr 22;15:17562848221090820. doi: 10.1177/17562848221090820. eCollection 2022. PMID 35480299